CLINICAL TRIAL: NCT06305780
Title: RECOVER-AUTONOMIC: A Platform Protocol for Evaluation of Interventions for Autonomic Dysfunction in Post-Acute Sequelae of SARS-CoV-2 Infection (PASC)
Brief Title: RECOVER-AUTONOMIC Platform Protocol
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kanecia Obie Zimmerman (Other)
Responsible Party: Sponsor-Investigator, Kanecia Obie Zimmerman, Associate Professor of Pediatrics, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00112597; OTA-21-015G (Other: NIH Grant to RTI; RTI subcontracting with DCRI)
Record Dates: First submitted 2024-03-04; First posted 2024-03-12 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Long COVID; Long Covid19; Long Covid-19
Keywords: PASC; POTS
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome | interventions — Immunoglobulins, Intravenous; Ivabradine

STUDY DESIGN:
Intervention Model Description: In each Appendix trial, each participant will be assigned with equal probability to one of the factorial combinations based on two factors: (1) a study intervention/control and (2) non-pharmacologic intervention/control if the participant is eligible for the study intervention.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IVIG (Experimental): In the IVIG study, randomization will be implemented with 1:1:1:1 allocation among the combination of IVIG/placebo and coordinated/ usual non-pharmacologic care. All participants will receive IVIG or placebo for 9 months (36 weeks) with a follow-up period for an additional 3 months (total study duration for 12 months). See NCT06305793 for additional details.
  Interventions: Drug: IVIG + Coordinated Care; Drug: IVIG Placebo + Coordinated Care; Drug: IVIG + Usual Care; Drug: IVIG Placebo + Usual Care
- Ivabradine (Experimental): In the ivabradine study, randomization will be implemented with 1:1:1:1 allocation among the combinations of ivabradine/placebo and coordinated/usual care. All participants receive either ivabradine or placebo for 3 months (12 weeks) with a follow-up period for an additional 3 months (total study duration of 6 months). See NCT06305806 for additional details.
  Interventions: Drug: Ivabradine + Coordinated Care; Drug: Ivabradine Placebo + Coordinated Care; Drug: Ivabradine + Usual Care; Drug: Ivabradine Placebo + Usual Care

INTERVENTIONS:
Drug: IVIG + Coordinated Care — Participants will receive IVIG for a duration of 9 months and coordinated non-pharmacologic care for a duration of 3 months, concurrent with IVIG administration. Coordinated non-pharmacologic care involves volume expansion through high salt diet, water intake, abdominal binder, exercise/rehabilitation, motivation, education, and assisted care through a care coordinator.
  Arms: IVIG
Drug: IVIG Placebo + Coordinated Care — Normal saline given intravenously will be the control (placebo) product. Blinding IV bag and tubing covers will be used for both IVIG and Placebo administration.
  Participants will receive IVIG placebo for a duration of 9 months and coordinated non-pharmacologic care for a duration of 3 months, concurrent with IVIG placebo administration. Coordinated non-pharmacologic care involves volume expansion through high salt diet, water intake, abdominal binder, exercise/rehabilitation, motivation, education, and assisted care through a care coordinator.
  Arms: IVIG
Drug: Ivabradine + Coordinated Care — Participants will receive Ivabradine for a duration of 3 months and coordinated non-pharmacologic care for a duration of 3 months, concurrent with ivabradine administration. Coordinated non-pharmacologic care involves volume expansion through high salt diet, water intake, abdominal binder, exercise/rehabilitation, motivation, education, and assisted care through care coordinator.
  Arms: Ivabradine
Drug: Ivabradine Placebo + Coordinated Care — The control (placebo) oral tablets will be similar to the study drug, ivabradine.
  The control packaging matches the packaging.
  Participants will receive Ivabradine placebo for a duration of 3 months and coordinated non-pharmacologic care for a duration of 3 months, concurrent with ivabradine placebo administration. Coordinated non-pharmacologic care involves volume expansion through high salt diet, water intake, abdominal binder, exercise/rehabilitation, feedback, nutrition counseling, motivation, education, and assisted care through care coordinator.
  Arms: Ivabradine
Drug: IVIG + Usual Care — Participants will receive IVIG for a duration of 9 months and usual non-pharmacologic care (control) for a duration of 3 months. This will be concurrent with scheduled IVIG administration.
  Arms: IVIG
Drug: IVIG Placebo + Usual Care — Normal saline given intravenously will be the control (placebo) product. The normal saline will be of similar formulation and appearance to IVIG.
  Participants will receive IVIG placebo for a duration of 9 months and usual non-pharmacologic care (control) for a duration of 3 months. This will be concurrent with scheduled IVIG placebo administration.
  Arms: IVIG
Drug: Ivabradine + Usual Care — Participants will receive Ivabradine for a duration of 3 months and usual non-pharmacologic care (control) for a duration of 3 months, concurrent with ivabradine administration.
  Arms: Ivabradine
Drug: Ivabradine Placebo + Usual Care — The control (placebo) oral tablets will be similar to the study drug, ivabradine.
  The control packaging matches the packaging.
  Participants will receive Ivabradine placebo for a duration of 3 months and usual non-pharmacologic care (control) for a duration of 3 months, concurrent with ivabradine placebo administration.
  Arms: Ivabradine

SUMMARY:
This study is a platform protocol designed to be flexible so that it is suitable for a wide range of settings within health care systems and in community settings where it can be integrated into COVID-19 programs and subsequent treatment plans.

This protocol is a prospective, multi-center, multi-arm, randomized, controlled platform trial evaluating various interventions for use in the treatment of autonomic dysfunction symptoms, including cardiovascular complications and postural orthostatic tachycardia syndrome (POTS), in PASC participants. The interventions tested will include non-pharmacologic care and pharmacologic therapies with study drugs.

DETAILED DESCRIPTION:
The hypothesis is that some of the autonomic dysfunction symptoms are immune-mediated, so immunotherapy and other applicable therapies will result in improvement in autonomic symptoms.

Interventions will be added to the platform protocol as appendices. Each appendix will leverage all elements of the platform protocol, with additional elements described in the individual appendix.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age at the time of enrollment
2. Previous suspected, probable, or confirmed SARS-CoV-2 infection, as defined by the Pan American Health Organization12ɸ ɸ Enrollment of participants with suspected or probable SARS-CoV-2 infection will only be allowed if they occurred before May 1, 2021 and be limited to no more than 10% of the total sample size per Study Drug Appendix. Refer to the Manual of Procedures (MOP) for details.

   Suspected case of SARS-CoV-2 infection - Three options, A through C:

   A. Meets the clinical OR epidemiological criteria.
   1. Clinical criteria: Acute onset of fever AND cough (influenza-like illness) OR Acute onset of ANY THREE OR MORE of the following signs or symptoms: fever, cough, general, weakness/fatigue, headache, myalgia, sore throat, coryza, dyspnea, nausea, diarrhea, anorexia.
   2. Epidemiological criteria: Contact of a probable or confirmed case or linked to a COVID-19 cluster; or B. Presents with acute respiratory infection with history of fever or measured fever of ≥ 38°C; and cough; with onset within the last 10 days; and who requires hospitalization); or C. Presents with no clinical signs or symptoms, NOR meeting epidemiologic criteria with a positive professional use or self-test SARS-CoV-2 antigen-Rapid Diagnostic Test.

   Probable case of SARS-CoV-2 infection, defined as meets clinical criteria above AND is a contact of a probable or confirmed case or is linked to a COVID-19 cluster.

   Confirmed case of SARS-CoV-2 infection - Two options, A through B:

   A. A person with a positive nucleic acid amplification test, regardless of clinical criteria OR epidemiological criteria; or B. Meeting clinical criteria AND/OR epidemiological criteria (See suspect case A). With a positive professional use or self-test SARS-CoV-2 Antigen-Rapid Diagnostic Test.
3. Moderate, self-identified autonomic symptoms (defined as COMPASS-31 >25) following a SARS-CoV-2 infection that has persisted for at least 12 weeks and is still present at the time of consent
4. OHQ/OIQ, question 1 score >2

Exclusion Criteria:

1. Known pregnancy, breast-feeding, or contemplating pregnancy during the study period
2. Known active acute SARS-CoV-2 infection ≤ 4 weeks from enrollment
3. Known renal failure (eGFR <20ml/1.73 m²)
4. Known atrial fibrillation or significant cardiac arrhythmia
5. Known cardiovascular conditions such as heart failure (Class 3-4), severe valvular disease, symptomatic ischemic coronary artery disease, revascularization for PAD/CAD within the past 6 months
6. Clinically significant atherosclerotic disease, defined as history of stroke or myocardial infarction or revascularization 6 months prior to enrollment and/or current symptomatic angina
7. Existing uncontrolled hypertension
8. History of significant hypercoagulability disorders
9. Active or recent thrombosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 381 (Actual)
Dates: Start 2024-03-11 (Actual); Primary Completion 2025-07-09 (Actual); Study Completion 2025-07-09 (Actual)

PRIMARY OUTCOMES:
Total number of participants enrolled in each Appendix | Baseline to End of Intervention (IVIG 9 months, Ivabradine 3 months)
  Total number of participants enrolled in each Appendix will be reported. Appendix-specific outcome measure data will be reported under the associated NCT#

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Granger, MD, Study Chair — Duke Clinical Research Institute; Cyndya Shibao, MD, Study Chair — Vanderbilt University Medical Center; Peter Novak, MD, Study Chair — Harvard; Pam Taub, MD, Study Chair — University of California, San Diego; Tae Chung, MD, Study Chair — Johns Hopkins University
Locations (50):
- United States (50):
  - East Alabama Medical Center - Appendix B Only, Opelika, Alabama
  - Center for Complex Neurology - Appendix A & B, Phoenix, Arizona
  - University of Arkansas for Medical Sciences - Appendix A & B, Little Rock, Arkansas
  - University of California San Diego - Appendix B Only, La Jolla, California
  - Cedars Sinai Medical Center - Appendix A & B, Los Angeles, California
  - Stanford University - Appendix B Only, Stanford, California
  - University of Colorado Anschutz Medical Campus Clinical and Translational Research Center (CTRC) - Appendix A & B, Aurora, Colorado
  - MedStar National Rehabilitation Hospital - Appendix B only, Washington D.C., District of Columbia
  - University of Florida Health - Appendix A & B, Gainesville, Florida
  - Lakeland Regional Medical Center - Appendix A & B, Lakeland, Florida
  - Innovation Clinical Trials Inc.- Appendix A & B, Palmetto Bay, Florida
  - Grady Memorial Hospital - Woodruff Memorial Research - Appendix A & B, Atlanta, Georgia
  - Morehouse School of Medicine - Appendix A & B, Atlanta, Georgia
  - Queens Medical Center - Appendix B Only, Honolulu, Hawaii
  - Rush University Medical Center - Appendix B Only, Chicago, Illinois
  - University of Illinois at Chicago - Appendix A & B, Chicago, Illinois
  - NorthShore University HealthSystem - Evanston Hospital - Appendix B Only, Evanston, Illinois
  - University of Iowa - Appendix A & B, Iowa City, Iowa
  - University of Kansas Medical Center CTSU Fairway - Appendix A & B, Fairway, Kansas
  - University of Kentucky Medical Center - Appendix A & B, Lexington, Kentucky
  - University Medical Center New Orleans - Appendix A & B, New Orleans, Louisiana
  - Johns Hopkins Hospital - Appendix A Only, Baltimore, Maryland
  - Brigham and Women's Hospital - Appendix A Only, Boston, Massachusetts
  - Henry Ford Hospital - Appendix A & B, Detroit, Michigan
  - Mayo Clinic - Appendix A & B, Rochester, Minnesota
  - University of Mississippi Medical Center - Appendix A & B, Jackson, Mississippi
  - Washington University School of Medicine - Appendix B Only, St Louis, Missouri
  - University at Buffalo - Appendix A & B, Buffalo, New York
  - St. Lawrence Health Medical Campus - Appendix A & B, Canton, New York
  - Columbia University Irving Medical Center - Appendix A & B, New York, New York
  - Stony Brook University Hospital - Appendix A & B, Stony Brook, New York
  - Montefiore Medical Center - Moses Campus - Appendix B, The Bronx, New York
  - Duke University Hospital - Appendix A & B, Durham, North Carolina
  - East Carolina University - Appendix B Only, Greenville, North Carolina
  - Cleveland Clinic - Appendix A & B, Cleveland, Ohio
  - University of Oklahoma Health Science Center - Oklahoma Clinical and Translational Science Institute - Appendix A & B, Oklahoma City, Oklahoma
  - Oregon Health and Science University - Appendix A & B, Portland, Oregon
  - Kent Hospital - Appendix A & B, Pawtucket, Rhode Island
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - National Neuromuscular Research Institute - Appendix A & B, Austin, Texas
  - Southwest Family Medicine Associates - Appendix A & B, Dallas, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - University of Texas Health Science Center at San Antonio - Appendix A & B, San Antonio, Texas
  - Bateman Horne Center - Appendix B Only, Salt Lake City, Utah
  - Vermont Lung Center, University of Vermont - Appendix B Only, Burlington, Vermont
  - University of Virginia Health System, University Hospital - Appendix A & B, Charlottesville, Virginia
  - Sentara Norfolk General Hospital - Appendix A & B, Norfolk, Virginia
  - Evergreen Hospital Medical Center - Appendix A & B, Kirkland, Washington
  - Providence Medical Research Center - Appendix A & B, Spokane, Washington
  - Marshall Health - University Physicians and Surgeons - Appendix A & B, Huntington, West Virginia

IPD SHARING:
Plan to Share IPD: No
The summary of results will be shared on the study website: https://recovercovid.org/

REFERENCES:
- See also: Related Info — http://recovercovid.org/

DOCUMENTS (1):
  • Informed Consent Form (2024-01-15): https://cdn.clinicaltrials.gov/large-docs/80/NCT06305780/ICF_000.pdf